CLINICAL TRIAL: NCT05197556
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Groups, Phase 2a Clinical Trial to Evaluate the Safety and Efficacy of HSG4112 in Overweight and Obese Patients Following 12 Weeks of Oral Treatment
Brief Title: A Study to Evaluate the Safety and Efficacy of HSG4112 in Overweight and Obese Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaceum (Industry)
Collaborators: Gangnam Severance Hospital (Other); Seoul National University Bundang Hospital (Other); Korea University Anam Hospital (Other); Seoul National University Hospital (Other); SMG-SNU Boramae Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSG4112-P2-01
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2022-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HSG4112 200 mg Multiple Dose (Experimental): Multiple oral dosing of HSG4112 200 mg for 12 weeks
  Interventions: Drug: HSG4112
- HSG4112 400 mg Multiple Dose (Experimental): Multiple oral dosing of HSG4112 400 mg for 12 weeks
  Interventions: Drug: HSG4112
- HSG4112 600 mg Multiple Dose (Experimental): Multiple oral dosing of HSG4112 600 mg for 12 weeks
  Interventions: Drug: HSG4112
- Placebo (Placebo Comparator): Multiple oral dosing of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSG4112 — Once-daily oral administration
  Other Names: 2-(8,8 dimethyl 2,3,4,8,9,10 hexahydropyrano[2,3 f]chromen 3 yl) 5 ethoxyphenol
  Arms: HSG4112 200 mg Multiple Dose; HSG4112 400 mg Multiple Dose; HSG4112 600 mg Multiple Dose
Drug: Placebo — Once-daily oral administration
  Arms: Placebo

SUMMARY:
1. Study Objective

   * To assess the effect of HSG4112 on body weight
   * To evaluate the safety and tolerability of HSG4112
2. Background

   Glaceum Inc. has evaluated the safety, tolerability, and pharmacokinetic/pharmacodynamic properties of HSG4112 in healthy subjects through its Phase 1 trials, and is planning to perform this Phase 2a trial to assess the safety and efficacy of HSG4112 in overweight and obese patients.
3. Number of Subjects

   This study is a Phase 2a clinical trial designed to evaluate the safety and efficacy of HSG4112 following multiple-dose administration. The subject sample size estimate for the primary efficacy endpoint was based on total body weight, and assumes repeated measurement of body weight occurs at Baseline and every 4 weeks thereafter during the 12-week treatment period. Based on similar weight loss studies with obesity drugs, the covariance matrix for body weight change over time is estimated as AR(1) (sigma = 3.07, rho = 0.9). Thus, with 20 subjects completing each treatment group, this study can detect a mean difference of 6 kg between HSG4112 and matching placebo treatments with 80% power, assuming a two-sided α-level of 0.05. Therefore, the target sample size for this study is 20 subjects/group.
4. Study Design and Protocol

This study is a randomized, double-blind, placebo-controlled, parallel-groups trial. Subjects deemed eligible to participate in this study based on the inclusion/exclusion criteria will be assigned a subject number and randomized to one of the 4 treatment groups - 1 group receiving placebo - in a 1:1:1:1 ratio. Subjects will be randomized to double-blind treatments and will receive a once-daily oral dose of the investigational product for 12 weeks according to the study protocol. Body weight and obesity/metabolism-related parameters will be evaluated to assess the efficacy of HSG4112. Assessments including measurement of vital signs, 12-lead ECG, clinical laboratory tests, pregnancy test, physical examination, and adverse event monitoring will be performed to evaluate the safety and tolerability of HSG4112. Blood samples will be collected for pharmacokinetic assessment and samples from subjects who have signed the consent form for the exploratory genetic research will undergo analysis to detect PON2 gene polymorphism.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form approved by the IRB before Screening.
2. 19 to 70 years, inclusive, at Screening.
3. BMI is 30 to 39.9 kg/m2, inclusive (obese), with or without comorbid conditions, or BMI is 27 to 29.9 kg/m2, inclusive (overweight), with at least 1 documented treated or untreated comorbid condition (e.g., hypertension, dyslipidemia, cardiovascular disease, glucose intolerance, sleep apnea). All comorbid conditions must be considered by the Investigator to be clinically stable.

   ☞ (BMI (kg/m2) = Weight (kg) / {Height (m)2})
4. Eligible females will be:

   * females of childbearing potential who are not pregnant, evidenced by a negative serum hCG pregnancy test at Screening
   * non-lactating, or
   * surgically sterile (defined as documented bilateral tubal ligation, bilateral tubal occlusion, bilateral oophorectomy, hysterectomy) or postmenopausal (defined as at least 12 months prior to Screening without menses with no alternative explanation for the absence of menses).
5. Eligible males should have no plans to have children up to 90 days following the last day of treatment.
6. A history of at least 1 unsuccessful weight loss attempt, per Investigator judgment.

Exclusion Criteria:

1. Clinically significant new illness, per Investigator judgment, in the 1 month before Screening and during the screening period.
2. Significant history or clinical manifestation of allergic reaction or hypersensitivity to the investigational product or any related drug compound.
3. Compliance with placebo self-administration is ≤80% during the 2-week single-blind placebo run-in period.
4. Weight loss >3% during the 2-week single-blind placebo run-in period.
5. Diabetes mellitus (type 1, type 2, or other). A remote history of gestational diabetes that has resolved is not exclusionary.
6. Previous or planned (for the duration of the study) bariatric surgery or device (i.e., gastric bypass, gastric banding, sleeve gastrectomy, gastric balloon, biliopancreatic diversion)
7. Anticipated surgery during the study that may interfere with study completion or compliance with the protocol.
8. Uncontrolled hypertension at Screening, defined as systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg. Subjects with uncontrolled hypertension at Screening may be re-screened >3 months following initiation or adjustment of antihypertensive therapy, if enrollment has not been closed.
9. Any of the following within 3 months of Screening: myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic attack, and cardiac arrhythmia requiring medical or surgical treatment.
10. Evidence of any other unstable or untreated clinically significant hepatic, renal, neurological, immunological, respiratory, endocrine, hematological, cardiovascular, psychiatric, or neoplastic disease, or disease that, based on Investigator's judgment, will make the subject inappropriate for the study.
11. Males with the following:

    * history of, or known cause of hypogonadism (e.g., treatment for prostate cancer)
    * history of infertility
    * Klinefelter's syndrome or Kallmann's syndrome
    * use of any medication within 6 months of Screening that can alter reproductive hormone levels, either as the intended effect or as a side effect, including: anabolic steroids, androstenedione, bicalutamide, cimetidine, dehydroepiandrosterone, diethylstilbestrol, other estrogens, dutasteride, finasteride, glucocorticoids (e.g., prednisone, cortisone, hydrocortisone, and decadron), oral ketoconazole, megestrol acetate, opiates (e.g., morphine, codeine, oxycodone, hydrocodone), spironolactone, testosterone or any androgen, and any medications for treating prostate cancer.
12. Major surgical procedure (intrathoracic, intracranial, intraperitoneal, liposuction) within 6 months of the Screening visit.
13. Congestive heart failure New York Heart Association class III and IV.
14. History of organ transplantation.
15. Screening TSH greater than 2x upper limit of normal. Subjects on L-thyroxine replacement must be on a stable dose for at least 6 weeks prior to Screening.
16. Hyperthyroidism (screening laboratory value TSH <lower limit of normal) and/or subjects taking methimazole, carbimazole, propylthiouracil, and/or beta-blockers for hyperthyroidism.
17. Fasting triglycerides >500 mg/dL at Screening. Subjects with elevated triglycerides at Screening may be re-screened >3 months after initiation or adjustment of lipid-lowering treatment, if study enrollment has not been closed.
18. Screening glycosylated hemoglobin (HbA1c) ≥6.5%.
19. Fasting plasma glucose ≥126 mg/dL.
20. Clinically significant abnormal hepatic (e.g., AST or ALT greater than 2.5x ULN, or total bilirubin greater than 2x ULN, unless documented Gilbert's syndrome) or renal function laboratory tests (e.g., glomerular filtration rate <60 mL/min).
21. Positive HBsAg, HCV Ab, HIV Ag/Ab, or VDRL at Screening.
22. Malignancy within 5 years of the Screening visit (except adequately treated cutaneous basal cell or squamous cell carcinoma).
23. All chronic medications (including but not limited to: antihypertensives, lipid-lowering drugs, cardiovascular drugs, antidepressants) must have been taken at a stable dose (and dosing interval) for at least 3 months prior to Screening.
24. Treatment within 1 month of the Screening visit with over-the-counter weight loss products or appetite suppressants (including herbal weight loss agents) or St. John's Wort, or within 3 months with an approved anti-obesity drug.
25. Recent (within 6 months of Screening) participation in any organized weight loss program (e.g., Juvis).
26. Treatment within 3 months of the Screening visit with systemic (i.e., oral or intravenous) steroids for ≥7-day duration.
27. Recent history (i.e., within 2 years prior to the Screening visit) of alcohol or drug abuse or a positive screen for drugs of abuse at Screening. Subjects with a positive drug screen may be eligible with approval from the Sponsor if the subject has a documented medical history requiring the need for chronic pain treatment and a documented concomitant medication resulting in a positive drug screen, and provided the subject is considered by the Investigator to be reliable to participate in the study.
28. Significant change in smoking habits within 3 months prior to Screening, as judged by the Investigator.
29. Participated in any other clinical study or bioequivalence study and was dosed with an investigaiontal product within 6 months prior to the first day of dosing, unless there is documentation that the subject received placebo.
30. Significant change in diet or level of physical activity within 1 month prior to Screening, based on Investigator's judgment.
31. Weight loss or gain of more than 5% within 3 months prior to the Screening visit by history or documented.
32. Unwilling, or whose partner is unwilling, to use a medically acceptable means of contraception during and for 90 days following completion/withdrawal of the study.

    ☞ Medically acceptable contraceptive methods include:
    * hormonal contraceptive
    * intrauterine device that has been proven highly effective, used by the subject or the subject's spouse/partner
    * physical contraception (male or female) used with chemical sterilization
    * surgical sterilization of the subject or the subject's partner (e.g., vasectomy, hysterectomy, tubal ligation, salpingectomy).
33. Subjects who, in the opinion of the Investigator, should not participate in in this study based on clinical laboratory test results or other reasons.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight (kg) from Baseline to End of Treatment | Day 1 to Week 12
  Change in body weight (kg)
Evaluation of Safety and Tolerability by Adverse Event Monitoring | Day -1 to 4 weeks following the last administration (Week 16)
  Number of adverse events, adverse drug reactions, serious adverse events, and suspected unexpected serious adverse reactions

SECONDARY OUTCOMES:
Percentage of Subjects with ≥5% Body Weight Loss from Baseline to End of Treatment | Day 1 to Week 12
  Percentage of subjects (%) with ≥5% body weight loss
Percentage of Subjects with ≥7% Body Weight Loss from Baseline to End of Treatment | Day 1 to Week 12
  Percentage of subjects (%) with ≥7% body weight loss
Percentage of Subjects with ≥10% Body Weight Loss from Baseline to End of Treatment | Day 1 to Week 12
  Percentage of subjects (%) with ≥10% body weight loss
Percent Change in Body Weight from Baseline to End of Treatment | Day 1 to Week 12
  Percent change (%) in body weight

CONTACTS AND LOCATIONS:
Overall Officials: Hyuktae Kwon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Min K, Oh B, Koo HY, Kim YH, Lee JW, Lee S, Kim Y, Kwon H. Effect of anti-obesity agent HSG4112 on overweight and obese patients following 12 weeks of oral treatment: a study protocol for a randomised, double-blind, placebo-controlled, parallel-group, phase 2a clinical trial. Front Pharmacol. 2023 Aug 24;14:1177539. doi: 10.3389/fphar.2023.1177539. eCollection 2023. PMID 37693914